CLINICAL TRIAL: NCT04236258
Title: A Randomized Controlled Trial Comparing Nifedipine and Enalapril in Medical Resources Used in the Postpartum Period
Brief Title: Comparing Nifedipine and Enalapril in Medical Resources Used in the Postpartum Period
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Thomas Frederick McElrath, M.D.,Ph.D., Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019P002981
Record Dates: First submitted 2020-01-16; First posted 2020-01-22 (Actual); Results first posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Hypertension in Pregnancy; Preeclampsia Severe; Gestational Hypertension; Postpartum Preeclampsia; Postpartum
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Enalapril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nifedipine (Active Comparator): This arm will be postpartum women with high blood pressure who need an antihypertensive and have been assigned to start nifedipine extended release 30 mg daily as their starting antihypertensive.
  Interventions: Drug: NIFEdipine ER
- Enalapril (Active Comparator): This arm will be postpartum women with high blood pressure who need an antihypertensive and have been assigned to start enalapril 10 mg daily as their starting antihypertensive.
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: NIFEdipine ER — Postpartum women with high blood pressure will be randomized to receive nifedipine extended release 30mg daily as their starting antihypertensive.
  Arms: Nifedipine
Drug: Enalapril — Postpartum women with high blood pressure will be randomized to receive enalapril 10 mg daily as their starting antihypertensive.
  Arms: Enalapril

SUMMARY:
This study evaluates whether nifedipine or enalapril is better at decreasing the amount of medical resources used in the postpartum period by women who have high blood pressure in pregnancy and the postpartum period. Half of participants will receive enalapril while the other half will receive enalapril. We will compare the two groups in the amount of medical resources used which we are defining as prolonged hospitalizations, unscheduled medical visits and/or hospital readmissions in the postpartum period.

DETAILED DESCRIPTION:
This is randomized controlled trial to investigate if enalapril is superior to nifedipine in terms of medical resources used in postpartum women with hypertension. These are both antihypertensives we commonly use in the postpartum period for women with hypertension in pregnancy but we do not know which medication works better at decreasing prolonged hospitalizations, the number of unscheduled medical visits and/or readmissions to the hospital.

Nifedipine is more traditionally used and well-validated by current medical literature. However, enalapril's mechanism of action is better suited to the dysregulation of blood pressure that can occur with hypertensive disorders of pregnancy. Therefore, we hypothesize that enalapril is superior to nifedipine in terms of medical resources used in the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of any hypertensive disorder of pregnancy/postpartum period or chronic hypertension
* provider wanting to initiate antihypertensive in the postpartum period
* the patient is not currently on >1 antihypertensive
* plans to receive postpartum care at the hospital or affiliated clinic

Exclusion Criteria:

* sustained pulse <60 or >120 BPM over four hours
* allergy to any of the antihypertensives
* creatinine greater than or equal to 1.5
* strict contraindication to any of the antihypertensives
* history of failed treatment with any of the antihypertensives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas McElrath, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available to other researchers for all primary and secondary outcomes as well as demographic data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available for approximately six months after the study's conclusion.
Access Criteria: Data access requests will be reviewed by the internal Institutional Review Board.

REFERENCES:
- [Derived] Yoselevsky EM, Seely EW, Celi AC, Robinson JN, McElrath TF. A randomized controlled trial comparing the efficacy of nifedipine and enalapril in the postpartum period. Am J Obstet Gynecol MFM. 2023 Dec;5(12):101178. doi: 10.1016/j.ajogmf.2023.101178. Epub 2023 Oct 6. PMID 37806651

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled 94 participants in the study.
Pre-assignment Details: We aimed for 90 participants as part of the protocol but ended up oversampling at 94 due to concern over potential drop out.
Period: Overall Study
Arm/Group | Nifedipine | Enalapril
Started | 47 | 47
Completed | 47 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nifedipine: Participants in the nifedipine group were assigned nifedipine ER 30mg daily as their initial antihypertensive.
- Enalapril: Participants in the nifedipine group were assigned enalapril 10mg daily as their initial antihypertensive.
- Total: Total of all reporting groups
Arm/Group | Nifedipine | Enalapril | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (6.3) | 32.4 (6.7) | 32.8 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants] — all participants in the study were female
  Participants
    Female | 47 | 47 | 94
    Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — This is self-identified race and/or ethnicity as derived from the electronic medical record.
  Participants
    Asian | 2 | 0 | 2
    Hispanic | 9 | 15 | 24
    Non-Hispanic Black | 11 | 17 | 28
    White | 25 | 15 | 40
Region of Enrollment [Number; unit: participants]
  United States | 47 | 47 | 94
Insurance [Count of Participants; unit: Participants]
  Public insurance | 15 | 21 | 36
  Private insurance | 32 | 26 | 58
Parity [Mean (Standard Deviation); unit: para] — number of live children a participant has
  para | 1.89 (1.6) | 1.85 (1.7) | 1.87 (1.7)
Twin gestation [Count of Participants; unit: Participants] | 9 | 2 | 11
Delivery type [Count of Participants; unit: Participants]
  Vaginal | 12 | 21 | 33
  Operative | 6 | 1 | 7
  Cesarean | 29 | 25 | 54
Gestational age at delivery [Mean (Standard Deviation); unit: weeks] | 36.6 (2.3) | 37.4 (2.9) | 36.9 (2.6)
Hypertensive diagnosis [Count of Participants; unit: Participants]
  Chronic | 3 | 3 | 6
  Gestational | 16 | 9 | 25
  Preeclampsia without severe features | 2 | 4 | 6
  Preeclampsia with severe features | 21 | 30 | 51
  Superimposed preeclampsia | 5 | 1 | 6
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.6 (8.0) | 35.2 (7.0) | 34.9 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Prolonged Hospitalization
Description: Participants who have any postpartum hospitalization that extends beyond the normal length of stay after delivery
Time Frame: up to six weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Enalapril
Number analyzed (Participants) | 47 | 47
Participants | 13 | 17

2. Primary Outcome: Unscheduled Clinic Appointment
Description: Participants who have any additional clinic appointments for any clinical reason in the postpartum period beyond the two appointments (around 1 week and 6 weeks postpartum) that are routinely scheduled
Time Frame: up to six weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Enalapril
Number analyzed (Participants) | 47 | 47
Participants | 19 | 17

3. Primary Outcome: Visit to Labor and Delivery Triage for Evaluation
Description: Participants who have any visit to triage on Labor and Delivery for evaluation in the postpartum period for any clinical reason
Time Frame: up to six weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Enalapril
Number analyzed (Participants) | 47 | 47
Participants | 13 | 17

4. Primary Outcome: Postpartum Readmission
Description: Participants who have any postpartum readmission after being discharged from the delivery hospitalization in the postpartum period
Time Frame: up to six weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Enalapril
Number analyzed (Participants) | 47 | 47
Participants | 3 | 4

5. Secondary Outcome: Time to Blood Pressure Control
Description: Time to sustained blood pressure control (defined as no need for changes to antihypertensive regimen for >24 hours)
Time Frame: up to six weeks postpartum
Measure: Mean (Standard Deviation); unit: days
Groups:
- Nifedipine: Patients who were initially randomized to nifedipine
- Enalapril: Patients who were initially randomized to enalapril
Arm/Group | Nifedipine | Enalapril
Number analyzed (Participants) | 47 | 47
days | 0.7 (1.0) | 1.9 (3.5)

6. Secondary Outcome: Number of Participants Who Needed for Additional Antihypertensives
Description: Any time a patient needs a second or third agent added to her antihypertensive regimen
Time Frame: up to six weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Enalapril
Number analyzed (Participants) | 47 | 47
Participants | 6 | 16

7. Secondary Outcome: Time to Discharge
Description: The days a patient stays in the hospital after delivery or after readmission for postpartum hypertension
Time Frame: up to six weeks postpartum
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nifedipine | Enalapril
Number analyzed (Participants) | 47 | 47
days | 3.2 (1.6) | 3.3 (1.7)

8. Secondary Outcome: Clinically Significant Hypotension or Hypertension
Description: Any time a patient became symptomatic from her blood pressure as noted by her providers
Time Frame: up to six weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Enalapril
Number analyzed (Participants) | 47 | 47
Participants | 0 | 0

9. Secondary Outcome: Creatinine Values at 1-2 Weeks After Discharge
Description: Creatinine measured at 1-2 weeks after discharge from the randomization hospitalization (not all study patients attended their appointments and had their blood drawn)
Time Frame: 1-2 weeks
Population: This is the population of participants who attended a 1-2 week clinic visit after discharge and had a creatinine level drawn
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nifedipine | Enalapril
Number analyzed (Participants) | 27 | 21
mg/dL | 0.68 (0.11) | 0.75 (0.17)

10. Secondary Outcome: Continued Need for Antihypertensive
Description: If a patient still needs the prescribed antihypertensives one week after discharge and six weeks after delivery to control her blood pressure as determined by her provider during her clinic visit
Time Frame: up to six weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Enalapril
Number analyzed (Participants) | 42 | 40
Participants | 41 | 36

11. Secondary Outcome: Number of Participants With Self-reported Side Effects Attributed to the Antihypertensive They Received
Description: A patient will complete a survey that will report any side effect the patient attributes to the antihypertension medication
Time Frame: up to six weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Enalapril
Number analyzed (Participants) | 13 | 13
Participants | 1 | 1

12. Secondary Outcome: Patient Self-reported Compliance With Their Antihypertensive Regimen
Description: The patient will complete a survey that self-assesses how compliant she has been with taking the prescribed antihypertensives ("difficulty remembering to take the medication")
Time Frame: up to six weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Enalapril
Number analyzed (Participants) | 13 | 13
Participants | 0 | 2

13. Secondary Outcome: Creatinine Level Around 6 Weeks After Delivery
Description: Creatinine level drawn at 6 week postpartum visit (not all study patients attended their appointments and had their blood drawn)
Time Frame: 6 weeks after delivery
Population: This is the population who attended their 6 week postpartum visit and had a creatinine level drawn at that time
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nifedipine | Enalapril
Number analyzed (Participants) | 12 | 13
mg/dL | 0.82 (0.15) | 0.88 (0.14)

ADVERSE EVENTS:
Time Frame: Data were collected for each patient over a period of 6 weeks after their delivery.
Arm/Group | Nifedipine | Enalapril
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47

LIMITATIONS AND CAVEATS:
The trial was conducted during the COVID pandemic which fundamentally changed the way patients interact with the medical system.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT04236258/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT04236258/SAP_001.pdf